CLINICAL TRIAL: NCT00003054
Title: Evaluation of Paclitaxel (Taxol) in the Treatment of Recurrent or Persistent Leiomyosarcoma of the Uterus
Brief Title: Paclitaxel in Treating Patients With Recurrent or Persistent Cancer of the Uterus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000065702; GOG-131C
Record Dates: First submitted 1999-11-01; First posted 2003-06-25 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Sarcoma
Keywords: recurrent uterine sarcoma; uterine leiomyosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients with recurrent or persistent cancer of the uterus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the antitumor activity of paclitaxel in patients with metastatic or persistent leiomyosarcoma of the uterus who have failed treatment protocols of higher priority. II. Determine the nature and degree of toxic effects of paclitaxel in this group of patients.

OUTLINE: Patients receive a continuous infusion of paclitaxel once every 3 weeks over 3 hours. Patients in complete remission, partial remission, or stable disease undergo at least 3 courses of paclitaxel. Paclitaxel continues until disease progression or adverse effects prohibit further treatment. All patients are followed until death.

PROJECTED ACCRUAL: This study anticipates an annual accrual of approximately 25 patients over 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or persistent uterine leiomyosarcoma that is refractory to curative therapy or established treatments Measurable disease required Must have failed local therapeutic measures and must be considered incurable Not eligible for GOG protocols of higher priority

PATIENT CHARACTERISTICS: Age: Not specified Performance status: GOG 0-3 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Granulocyte count at least 1,500/mm3 Hepatic: Bilirubin no greater than 1.5 times normal SGOT and alkaline phosphatase no greater than 3 times normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No unstable angina within 6 months OR No myocardial infarction within 6 months Abnormal cardiac condition (e.g., bundle branch block, heart block) allowed if stable for 6 months Other: No significant infection No concomitant malignancy other than nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: At least 3 weeks since prior therapy to malignant tumor Biologic therapy: Not specified Chemotherapy: Recovery from prior chemotherapy required No more than 1 prior chemotherapy regimen allowed No prior paclitaxel No prior chemotherapy for any malignancy from which the patient is disease-free for at least 5 years Endocrine therapy: Not specified Radiotherapy: Recovery from prior radiation therapy required No prior radiation therapy for any malignancy from which the patient is disease-free for at least 5 years Surgery: Recovery from prior surgery required

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-08; Primary Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald G. Gallup, MD, Study Chair — Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center
Locations (65):
- United States (64):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Medical College of Georgia Comprehensive Cancer Center, Augusta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Medicine Branch, Bethesda, Maryland
  - Radiation Oncology Branch, Bethesda, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Brookview Research, Inc., Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - St. Francis Hospital/Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- NCIC-Clinical Trials Group, Kingston, Ontario, Canada

REFERENCES:
- [Result] Gallup DG, Blessing JA, Andersen W, Morgan MA; Gynecologic Oncology Group Study. Evaluation of paclitaxel in previously treated leiomyosarcoma of the uterus: a gynecologic oncology group study. Gynecol Oncol. 2003 Apr;89(1):48-51. doi: 10.1016/s0090-8258(02)00136-1. PMID 12694653